CLINICAL TRIAL: NCT05079516
Title: Neural Basis of Sensory Learning: Brain Regions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hannah Justine Block, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 12517; R01NS112367-01A1 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-10-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Basic Science

STUDY DESIGN:
Intervention Model Description: The study includes two experiments. Experiment 1 includes Arms 1-3, and Experiment 2 includes Arms 4-7. Arm assignment will be random within each experiment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Primary motor cortex--Exp 1 (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over primary motor cortex.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Somatosensory cortex--Exp 1 (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over primary somatosensory cortex.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Vertex sham--Exp 1 (Sham Comparator): Sham theta burst transcranial magnetic stimulation (cTBS) will be applied over the vertex.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Anterior superior parietal lobule--Exp 2 (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over Anterior superior parietal lobule.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Ventral premotor cortex--Exp 2 (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over Ventral premotor cortex.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Cerebellar cortex--Exp 2 (Experimental): Theta burst transcranial magnetic stimulation (cTBS) will be applied over cerebellar cortex.
  Interventions: Other: Theta burst transcranial magnetic stimulation
- Vertex sham--Exp 2 (Sham Comparator): Sham theta burst transcranial magnetic stimulation (cTBS) will be applied over the vertex.
  Interventions: Other: Theta burst transcranial magnetic stimulation

INTERVENTIONS:
Other: Theta burst transcranial magnetic stimulation — Real or sham continuous theta burst TMS (cTBS) will be delivered to a location on the head, determined by randomized group assignment. cTBS consists of 600 low-intensity TMS pulses delivered over 40 seconds in a pattern of 50 Hz triplets delivered at 5 Hz.

SUMMARY:
The purpose of this study is to understand how the sensory and motor areas of the brain work together to keep a person's hand movements accurate (sensorimotor learning). The investigators hope this information may be useful one day to improve rehabilitation techniques in patients with brain lesions.

DETAILED DESCRIPTION:
To make accurate movements, the brain needs to compensate for the frequent changes in the environment one experiences (lighting conditions, slippery floors, etc). For example, when one reaches to grab an object underwater, there are significant challenges the brain must overcome. Water is more viscous than air, so motor planning must take the increased resistance into account. In addition, light is bent by water, so one sees the underwater hand in a different location from where one feels it with body position sense (proprioception, from sensors in the joints and muscles). While initially movement errors occur in a situation like this, a healthy person quickly learns to compensate. This compensation can take different forms. The brain can shift the proprioceptive estimate closer to the visual estimate of hand position or vice versa (sensory realignment), or the brain can compensate for any movement errors by altering the motor commands to the arm (motor adaptation).

Failure to compensate for such changes results in inaccurate movement, raising the potential for accidents and injuries, but how the healthy brain carries out these functions, and how they could be strengthened in populations with sensory and motor deficits (e.g. stroke), is unknown. With greater understanding of these processes in the healthy brain, it may one day be possible to develop rehabilitation strategies that target a patient's unique mix of sensory and motor deficits.

A robust way to identify whether a brain region plays a role in a behavior is to temporarily modulate its excitability in healthy people using non-invasive brain stimulation. This is commonly done in research with a short sequence of low-intensity transcranial magnetic stimulation (TMS), also known as repetitive TMS (rTMS). rTMS is used clinically to treat conditions such as depression and is considered very low risk provided the generally-accepted screening criteria are met. In the research setting, this technique is widely used not only in healthy adults (as in this study) but also in children and people with concussion, stroke, Parkinson's disease, and more.

In separate groups of subjects, the investigators will use a 40-second sequence of rTMS called continuous theta burst stimulation (cTBS) over one of several brain regions of interest before the subject performs a reaching task known to involve sensory realignment (learning). If performance of the task is affected by cTBS for a given group (relative to the sham, or control, group), it means that brain region plays some role in that type of reaching task.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must be between the ages of 18-45 years old and right-handed. Aging has been shown to affect the morphology of sensory and motor nerves, conduction velocities of nerves, and number of motor neurons in the spinal cord; to avoid these confounding factors we will only examine younger-to middle-aged adults.
* There are differences in cortical function and corticospinal projections such that testing the right arm of a right-handed individual is not necessarily equivalent to testing the left arm of a left-handed individual. To eliminate this confound, we will only test right-handed individuals. All these factors will be determined with the initial screening questions.
* Covid has been found to have neurological effects in some people, but mostly the effects on sensorimotor control and neurophysiology are unknown. So we want to reduce the chances of inadvertently testing subjects who have covid. We will therefore only include individuals who are fully vaccinated (2+ weeks past their final vaccine dose) or have a negative Covid test within 4 days of testing. We will further only include individuals who report being free of Covid symptoms in week preceding testing.

Exclusion Criteria:

1. Determined with initial screening questions, pre-enrollment:

   Potential subjects will be excluded for current vision problems, other than needing glasses or contacts. Subjects will also be excluded if they currently suffer from frequent severe headaches, glaucoma, heart or respiratory disease, hypertension, psychiatric conditions, or learning or attention conditions. They will also be excluded for current or past: visual, hearing, or balance impairments; stroke, seizure/epilepsy (including family history), or severe head trauma; fainting; or diabetes. Subjects will be excluded for metal implants in the head other than titanium; cochlear implants; implanted neurostimulator; cardiac pacemaker; intracardiac lines; or a medication infusion device. Because TMS does not penetrate deeply into the head, we cannot test subjects whose hair does not permit contact between the TMS coil and the scalp. We will therefore exclude subjects with dreadlocks, weaves, or hair extensions. To protect the data from extraneous peripheral influences, we will also exclude subjects who have had serious injury to the bones, joints, or muscles of either hand or arm, and have not fully recovered. For the purpose of this study, "fully recovered" means they no longer notice any pain, weakness, or loss of sensation in the injured area, and have no mobility limitations.

   For the validity of our data, we will exclude subjects taking medications or drugs that are known to affect cortical excitability and possibly seizure risk in an rTMS study. These medications/drugs are (Rossi et al., 2009): imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, sympathomimetics.
2. Determined on each day of TMS testing:

   Potential subjects will be invited to reschedule if they would otherwise be eligible (according to the initial screening), but the day of testing have drunk more than 3 units of alcohol or taken other recreational drugs in the 24 hour period prior to testing; have had more than 3 cups of coffee in the last hour; are sleep deprived (<4 hours sleep the previous night); or have participated in another brain stimulation experiment the same day. These are standard in the TMS literature to protect the validity of the data and keep seizure risk minimal. In addition, we will invite invite subjects to reschedule if they have any of the common Covid symptoms within the last week and if they haven't been fully vaccinated or obtained a negative Covid test within the past 4 days. If they don't believe they can meet these criteria on another date, they will be excluded.
3. Determined during the Familiarization session.

After giving their consent, participants may be excluded during or after the familiarization session if they are unable to perform the reaching task or follow instructions, or if their TMS stimulation parameters cannot be reliably determined by the experimenter, or if TMS is not well tolerated.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Realignment | 1 day
  Measured by comparing where the subject points on a touchscreen when indicating perceived position of visual and proprioceptive targets early vs. late in the behavioral task.

SECONDARY OUTCOMES:
Visuo-proprioceptive weighting | 1 day
  The degree to which participant relies on vision vs. proprioception when both are available. Measured by comparing where the subject points on a touchscreen when indicating perceived position of visual vs. proprioceptive targets.
Target hand reaching | 1 day.
  Location participant points at with no performance feedback.
Target estimation variance | 1 day
  Variance with which participant estimate visual and proprioceptive target positions. Computed from where subjects point at targets on a touchscreen.
Motor cortex excitability (arms 1-3) | 1 day
  mean motor evoked potential amplitude at SI1mV (stimulus intensity that elicits 1 mV response). Measured pre- and post-cTBS in Arms 1-3 only.
Tactile sensitivity (arms 1-3) | 1 day
  Two-point discrimination threshold on the target index fingertip. Measured pre- and post-cTBS in Arms 1-3 only.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah J Block, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results published in peer-reviewed journals will be shared. Only de-identified data will be shared.
Supporting Information: Analytic Code
Time Frame: The data will become available when group results are published in peer-reviewed journals.
Access Criteria: Data will be available on www.osf.io for anyone who wishes to download it. The relevant osf registry will be cited in the peer-reviewed publication so that interested readers can find it.